CLINICAL TRIAL: NCT05916365
Title: A 2-year Open-label Extension Study to Assess the Long-term Safety and Efficacy of Lebrikizumab in Adult and Adolescent Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Long-term Safety and Efficacy of Lebrikizumab in Adult and Adolescent Participant With Moderate-to-Severe Atopic Dermatitis
Acronym: ADlong
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-17923-32; 2022-502575-30-00 (Other: EU CTIS)
Record Dates: First submitted 2023-05-30; First posted 2023-06-23 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis
Keywords: Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis | interventions — lebrikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lebrikizumab (Experimental): Adult and adolescent participants (12 to less than [<] 18 years and weighing greater than or equal to [>=] 40 kilogram [kg]) with moderate-to-severe AD will receive lebrikizumab 250 milligrams (mg) subcutaneous (SC) injection via pre-filled syringe (PFS) for every fourth week (Q4W) for up to Week 104. If participants response is below EASI50 at any visit, lebrikizumab dosing frequency may be increased to every two weeks (Q2W) at any time during the course of the study; thereafter, lebrikizumab Q4W dosing may be resumed at the Investigator's discretion. Lebrikizumab will be administered up to Week 106 for participants who continue Q2W dosing, and these participants will undergo a safety follow-up assessment at Week 110.
  Interventions: Biological: Lebrikizumab

INTERVENTIONS:
Biological: Lebrikizumab — Lebrikizumab solution for injection administered subcutaneously

SUMMARY:
The main purpose of the study is to assess the long-term tolerability and effectiveness of lebrikizumab in adult and adolescent participants with moderate-to-severe atopic dermatitis (AD). Participants who complete the last assessment visit in ADjoin (Week 100) will be offered the opportunity to enroll in this extension study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who completed treatment with lebrikizumab in ADjoin and their last participant assessment visit (Week 100) in that study.
2. For WOCBP: agree to remain abstinent (refrain from heterosexual intercourse) or use a highly effective contraceptive method during the treatment period and for at least 4 weeks after the last dose of lebrikizumab.

   NOTE: A WOCBP is defined as a postmenarcheal female, who has not reached a postmenopausal state (>=12 continuous months of amenorrhea with no identified cause other than menopause) and has not undergone surgical sterilization (removal of ovaries, fallopian tubes, and/or uterus).

   NOTE: The following are highly effective contraceptive methods: combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) associated with inhibition of ovulation, progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, bilateral tubal ligation, vasectomized partner, or sexual abstinence. In the context of this protocol, sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post ovulation methods) and withdrawal are not acceptable methods of contraception.
3. Ability to understand the purpose and risks of the trial, willingness and ability to comply with the protocol and provide written informed consent/assent in accordance with institutional and regulatory guidelines.
4. Capable of giving signed informed consent/assent as described in which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Participants who, having participated in ADjoin, had their last lebrikizumab dose administered in a window longer than 8 weeks prior to the Baseline Visit in the current study.
2. Participants who, during their participation in the parent trial or ADjoin, developed an SAE or a severe AE that was deemed related to lebrikizumab, which in the opinion of the Investigator or of the medical monitor could indicate that continued treatment with lebrikizumab may present an unreasonable risk for the participant.
3. Conditions in the parent study or ADjoin consistent with protocol-defined criteria for permanent study drug discontinuation, if deemed related to lebrikizumab or led to Investigator or Sponsor-initiated withdrawal of participant from the study (e.g., non-compliance, inability to complete study assessments, etc.).
4. Treatment with a live (attenuated) vaccine from the time of last lebrikizumab dose in ADjoin prior to enrolment in the current study or planned during the study.
5. Use of a prohibited medication from the time of last lebrikizumab dose in ADjoin prior to enrolment in the current study or planned during the study.
6. Pregnant or breastfeeding women, and women planning to become pregnant or breastfeed during the study and for at least 4 weeks after the last dose of lebrikizumab.
7. Severe concomitant illness(es) that in the Investigator's judgment would adversely affect the participant's participation in the study. Any other medical or psychological condition that in the opinion of the Investigator may suggest a new and/or insufficiently understood disease, may present an unreasonable risk to the study patient because of his/her participation in this clinical trial, may make participant's participation unreliable, or may interfere with study assessments.
8. Any other conditions that, in the Investigator's opinion, might indicate the participant to be unsuitable for the trial.
9. Participant who is an employee or relative of an employee at the research site or Almirall.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of the Participants who will Discontinue from Study Treatment due to Treatment-emergent Adverse Events (TEAEs) | Baseline up to Week 110

SECONDARY OUTCOMES:
Percentage of Participants with Eczema Area and Severity Index (EASI) 50, EASI 75, and EASI 90 (>=50%, >=75%, and >=90%) Reduction in EASI Scores | Baseline up to Week 108
  The EASI is used to assess the severity and extent of AD; it is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and or extensive disease. EASI 50 is defined as 50% reduction from baseline in the EASI score. EASI 75 is defined as 75% reduction from baseline in the EASI score. EASI 90 is defined as 90% reduction from baseline in the EASI score.
Percentage Change from Baseline of Parent study in EASI Score | Baseline up to Week 108
  The EASI is used to assess the severity and extent of AD; it is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and or extensive disease. Baseline (i.e., prior to first study drug administration) is defined for the parent studies, J2T-DM-KGAB (ADvocate-1), J2TDM-KGAC (ADvocate-2), J2T-DM-KGAD (ADhere), and J2T-DM-KGAE (ADore).
Percentage of Participants with EASI Score <=7 | Baseline up to Week 108
  The EASI is used to assess the severity and extent of AD; it is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and or extensive disease. Baseline (i.e., prior to first study drug administration) is defined for the parent studies, J2T-DM-KGAB (ADvocate-1), J2TDM-KGAC (ADvocate-2), J2T-DM-KGAD (ADhere), and J2T-DM-KGAE (ADore).
Percentage of Participants Achieving Investigator Global Assessment (IGA) Score of 0 or 1 | Baseline up to Week 108
  The IGA is an instrument used to globally rate the severity of the participants AD. It is based on a 5-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate) and 4 (severe), and a score is selected using descriptors that best describe the overall appearance of the lesions at a given time point. The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Percentage of Participants Achieving Pruritus Numeric Rating Score (NRS) <= 4 | Baseline up to Week 108
  The Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours, with 0 indicating "No itch," and 10 indicating "Worst itch imaginable.
Percentage Change From Baseline of Parent Study in Body Surface Area (BSA) Involvement | Baseline to Week 108
  BSA affected by AD will be assessed for 4 separate body regions: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). BSA was calculated using the participant's palm using the 1% rule, 1 palm was equivalent to 1% with estimates of the number of palms it takes to cover the affected AD area. Maximum number of palms were 10 palms for head and neck (10%), 20 palms for upper extremities (20%), 30 palms for trunk, including axilla and groin (30%), 40 palms for lower extremities, including buttocks (40%). %BSA for a body region was calculated as = total number of palms in a body region * % surface area equivalent to 1 palm. Overall percent BSA of all 4 body regions ranges from 0% to 100 % with higher values represent greater severity of AD. Baseline (i.e., prior to first study drug administration) is defined for the parent studies, J2T-DM-KGAB (ADvocate-1), J2TDM-KGAC (ADvocate-2), J2T-DM-KGAD (ADhere), and J2T-DM-KGAE (ADore).
Proportion of Participants with Topical Corticosteroids (TCS)-free Days | Baseline up to Week 108
  Proportion of participants TCS- free days will be reported.
Percentage of Participants with DLQI/CDLQI Score <=5 | Baseline up to Week 108
  The DLQI is a 10-item validated questionnaire cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0 to 3 ("not at all," "a little", "a lot," and "very much"), giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. The CDLQI is validated from adolescents younger than age of 16 years, which is based on a set of 10 questions different from those of the DLQI. Each question is scored from 0 to 3, giving a possible total score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
Percentage of Participants Achieving at Least a 4-point Improvement from Baseline of Parent Study Dermatology Quality of Life Index/ Children's Dermatology Quality of Life Index (DLQI/CDLQI) | Baseline to Week 108
  The DLQI is a 10-item validated questionnaire cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0 to 3 ("not at all," "a little", "a lot," and "very much"), giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. The CDLQI is validated from adolescents younger than age of 16 years, which is based on a set of 10 questions different from those of the DLQI. Each question is scored from 0 to 3, giving a possible total score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life). Baseline (i.e., prior to first study drug administration) is defined for the parent studies, J2T-DM-KGAB (ADvocate-1), J2TDM-KGAC (ADvocate-2), J2T-DM-KGAD (ADhere), and J2T-DM-KGAE (ADore).

OTHER OUTCOMES:
Number of Participants with TEAEs, Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) | Baseline up to Week 110

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Stjepanovic, Principal Investigator — Almirall, S.A.
Locations (32):
- Germany (12):
  - Investigator Site 7, Darmstadt, Hesse
  - Investigator Site 8, Frankfurt am Main, Hesse
  - Investigator Site 10, Bad Bentheim, Lower Saxony
  - Investigator Site 9, Osnabrück, Lower Saxony
  - Investigator Site 11, Münster, North Rhine-Westphalia
  - Investigator Site 12, Leipzig, Saxony
  - Investigator Site 1, Augsburg
  - Investigator Site 2, Berlin
  - Investigator Site 3, Berlin
  - Investigator Site 4, Dresden
  - Investigator Site 5, Hamburg
  - Investigator Site 6, Hamburg
- Poland (20):
  - Investigator Site 26, Krakow, Lesser Poland Voivodeship
  - Investigator Site 25, Krakow, Lesser Poland Voivodeship
  - Investigator Site 23, Wroclaw, Lower Silesian Voivodeship
  - Investigator Site 28, Warsaw, Masovian Voivodeship
  - Investigator Site 27, Warsaw, Masovian Voivodeship
  - Investigator Site 31, Iwonicz-Zdrój, Podkarpackie Voivodeship
  - Investigator Site 32, Katowice, Silesian Voivodeship
  - Investigator Site 29, Ossy, Silesian Voivodeship
  - Investigator Site 30, Gdansk, Woj. Pomorskie
  - Investigator Site 13, Gdansk
  - Investigator Site 14, Katowice
  - Investigator Site 15, Kielce
  - Investigator Site 16, Lublin
  - Investigator Site 17, Poznan
  - Investigator Site 18, Rzeszów
  - Investigator Site 19, Szczecin
  - Investigator Site 20, Tarnów
  - Investigator Site 21, Warsaw
  - Investigator Site 22, Wroclaw
  - Investigator Site 24, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Undecided